CLINICAL TRIAL: NCT01096355
Title: A Phase I Study of Various Administration Schedules of RO4929097 With Multi-parameter Assessment (Biomarkers, Pharmacokinetics, Pharmacodynamics) in Patients With Advanced Solid Cancers
Brief Title: Gamma-Secretase Inhibitor RO4929097 in Treating Patients With Metastatic or Unresectable Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01550; NCI-2011-01550 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000666959; PMH-PJC-003; PJC-003 (Other: University Health Network-Princess Margaret Hospital); 8501 (Other: CTEP); U01CA132123 (NIH)
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2013-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide; Pharmacogenomic Testing

ARMS (6):
- Group A (Experimental): Patients receive oral gamma-secretase inhibitor RO4929097 once daily on days 1-3 and 8-10.
  Treatment in all groups repeats every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsies at baseline and between days 15 and 22 in the first course of treatment. Plasma samples are collected periodically for pharmacokinetic, pharmacodynamic, and pharmacogenomic analysis and to assess levels of adipsin and markers of angiogenesis.
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Other: diagnostic laboratory biomarker analysis; Other: pharmacogenomic studies; Other: pharmacological study
- Group B (Experimental): Patients receive oral RO4929097 once daily on days 1-7.
  Treatment in all groups repeats every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsies at baseline and between days 15 and 22 in the first course of treatment. Plasma samples are collected periodically for pharmacokinetic, pharmacodynamic, and pharmacogenomic analysis and to assess levels of adipsin and markers of angiogenesis.
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Other: diagnostic laboratory biomarker analysis; Other: pharmacogenomic studies; Other: pharmacological study
- Group C (Experimental): Patients receive oral RO4929097 once daily on days 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, and 21.
  Treatment in all groups repeats every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsies at baseline and between days 15 and 22 in the first course of treatment. Plasma samples are collected periodically for pharmacokinetic, pharmacodynamic, and pharmacogenomic analysis and to assess levels of adipsin and markers of angiogenesis.
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Other: diagnostic laboratory biomarker analysis; Other: pharmacogenomic studies; Other: pharmacological study
- Group D (Experimental): Patients receive oral RO4929097 once daily on days 1, 8, and 15.
  Treatment in all groups repeats every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsies at baseline and between days 15 and 22 in the first course of treatment. Plasma samples are collected periodically for pharmacokinetic, pharmacodynamic, and pharmacogenomic analysis and to assess levels of adipsin and markers of angiogenesis.
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Other: diagnostic laboratory biomarker analysis; Other: pharmacogenomic studies; Other: pharmacological study
- Group E (Experimental): Patients receive oral RO4929097 once daily on days 1, 4, 8, 11, 15, and 18.
  Treatment in all groups repeats every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsies at baseline and between days 15 and 22 in the first course of treatment. Plasma samples are collected periodically for pharmacokinetic, pharmacodynamic, and pharmacogenomic analysis and to assess levels of adipsin and markers of angiogenesis.
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Other: diagnostic laboratory biomarker analysis; Other: pharmacogenomic studies; Other: pharmacological study
- Group F (Experimental): Patients receive oral RO4929097 once daily days 1-5, 8-12, and 15-19.
  Treatment in all groups repeats every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsies at baseline and between days 15 and 22 in the first course of treatment. Plasma samples are collected periodically for pharmacokinetic, pharmacodynamic, and pharmacogenomic analysis and to assess levels of adipsin and markers of angiogenesis.
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Other: diagnostic laboratory biomarker analysis; Other: pharmacogenomic studies; Other: pharmacological study

INTERVENTIONS:
Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097
  Other Names: R4733; RO4929097
Other: diagnostic laboratory biomarker analysis
Other: pharmacogenomic studies
  Other Names: Pharmacogenomic Study
Other: pharmacological study
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects, best way to give, and best dose of gamma-secretase inhibitor RO4929097 in treating patients with metastatic or unresectable solid malignancies. Enzyme inhibitors, such as gamma-secretase inhibitor RO4929097, may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety profile of 6 different administration schedules of gamma-secretase inhibitor RO4929097 in patients with advanced solid malignancies.

SECONDARY OBJECTIVES:

I. To determine pharmacokinetic (PK) parameters of gamma-secretase inhibitor RO4929097 administered using 6 different administration schedules.

II. To assess the preliminary antitumor activity of gamma-secretase inhibitor RO4929097 in these patients.

TERTIARY OBJECTIVES:

I. To assess the pharmacodynamic (PD) effects of gamma-secretase inhibitor RO4929097 on Notch signaling pathway in tumor and surrogate tissues, as well as soluble markers of angiogenesis in plasma, when administered using 6 different dosing schedules. (Exploratory) II. To evaluate the relationship between PK and PD effects in an attempt to define the optimal biological dosing schedule (OBDS) that can provide a sustained inhibition of Notch signaling pathway over time with a tolerable toxicity profile. (Exploratory) III. To correlate inhibition of Notch signaling pathway measured in tumor and surrogate tissues with preliminary antitumor activity and assess the potential clinical predictive value of OBDS as defined above. (Exploratory) IV. To assess the effect of the various pharmacogenomic polymorphisms of the cytochrome P450 pathway on PK and PD parameters. (Exploratory)

OUTLINE: This is a multicenter, dose-escalation study. Patients are assigned to 1 of 6 dose schedules.

GROUP A: Patients receive oral gamma-secretase inhibitor RO4929097 once daily on days 1-3 and 8-10.

GROUP B: Patients receive oral RO4929097 once daily on days 1-7.

GROUP C: Patients receive oral RO4929097 once daily on days 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, and 21.

GROUP D: Patients receive oral RO4929097 once daily on days 1, 8, and 15.

GROUP E: Patients receive oral RO4929097 once daily on days 1, 4, 8, 11, 15, and 18.

GROUP F: Patients receive oral RO4929097 once daily days 1-5, 8-12, and 15-19.

Treatment in all groups repeats every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsies at baseline and between days 15 and 22 in the first course of treatment. Plasma samples are collected periodically for pharmacokinetic, pharmacodynamic, and pharmacogenomic analysis and to assess levels of adipsin and markers of angiogenesis.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid malignancy

  * Metastatic or unresectable disease
  * Standard curative or palliative measures do not exist or are no longer effective
* Measurable disease, defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan
* No known brain metastases
* ECOG performance status (PS) 0-1 (Karnofsky PS 70-100%)
* Life expectancy > 12 weeks
* Leukocytes ≥ 3,000/mm^3
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Total bilirubin normal
* AST/ALT ≤ 2.5 times upper limit of normal
* Serum creatinine normal OR creatinine clearance ≥ 60 mL/min
* No uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia, or hypokalemia, defined as < lower limit of normal despite adequate electrolyte supplementation
* QTc ≤ 450 msec in males and a QTc ≤ 470 in females, as measured by ECG using Bazett's formula
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 forms of contraception (i.e., barrier contraception and 1 other method of contraception) for ≥ 4 weeks before, during, and for ≥ 12 months after completion of study treatment
* Willing to undergo 2 tumor biopsies (unless medically contraindicated)
* Able to swallow medication
* No malabsorption syndrome or other condition that would interfere with intestinal absorption
* No diarrhea ≥ grade 2 not under control with standard antidiarrhea medications
* No uncontrolled concurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia other than chronic, stable atrial fibrillation
  * Psychiatric illness or social situations that would limit compliance with study requirements
* No history of risk factors for QT interval prolongation including, but not limited to, a family or personal history of any of the following:

  * Long QT syndrome
  * A history of torsades de pointes
  * Recurrent syncope without known etiology
  * Sudden unexpected death
* Female patients may not donate ova during or after study treatment
* No blood donation during and for ≥ 12 months after completion of study treatment
* No serologic positivity for hepatitis A, B, or C; history of liver disease; or other forms of hepatitis or cirrhosis
* No HIV-positive patients on combination antiretroviral therapy
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to gamma-secretase inhibitor RO4929097 or other agents used in this study
* No other concurrent agents or therapies administered with the intent to treat the patient's malignancy
* No prior gamma-secretase inhibitors
* Any number of prior treatment regimens allowed
* At least 4 weeks since prior radiotherapy or systemic therapy (6 weeks for prior carmustine or mitomycin C)

  * Exceptions may be made for low-dose, nonmyelosuppressive radiotherapy for symptomatic palliation
* Recovered from the adverse events due to prior therapy to < CTCAE grade 2 (except alopecia)
* No other concurrent investigational agents
* No concurrent medications with narrow therapeutic indices that are metabolized by cytochrome P450, including warfarin sodium (Coumadin®)
* No concurrent medications that are strong inducers/inhibitors or substrates of CYP3A4
* No concurrent medications or food that may interfere with the metabolism of gamma-secretase inhibitor RO4929097 including ketoconazole, grapefruit, or grapefruit juice
* No antiarrhythmics or other concurrent medications with known potential to prolong QT interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-02; Primary Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Safety profile of six different administration schedules of RO4929097 | Up to 4 weeks

SECONDARY OUTCOMES:
Determination of pharmacokinetic profiles of various administration schedules | Up to 4 weeks
Preliminary antitumor activity of RO4929097 assessed using RECIST 1.1 criteria | Up to 4 weeks
Pharmacokinetic (PK) parameters of RO4929097 administered using six different dosing schedules | Up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (3):
- Canada (3):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario